CLINICAL TRIAL: NCT00561327
Title: PPARgamma Activation by Losartan in Hypertensive Patients: The Importance of Losartan-Metabolites
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: German Heart Institute (Other)
Collaborators: Charite University, Berlin, Germany (Other); Merck Sharp & Dohme LLC (Industry)
Other Study IDs: P2132V1
Record Dates: First submitted 2007-11-16; First posted 2007-11-20 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-07

CONDITIONS: Hypertension
Keywords: hypertension; angiotensin receptor blockers; peroxisome proliferator activated receptor gamma
MeSH Terms: conditions — Hypertension | interventions — Losartan

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: Patients chronically treated with drug losartan
  Interventions: Drug: losartan
- B: Patients not chronically treated with losartan

INTERVENTIONS:
Drug: losartan — Daily treated with losartan 100mg for at least the past 2 months (retrospective, no new drug treatment/ intervention)
  Groups: A

SUMMARY:
The purpose of this study is to determine whether losartan metabolites are effective in inducing PPARγ target genes in monocytes in losartan-treated patients.

DETAILED DESCRIPTION:
The losartan metabolite EXP3179 potently induces the activity of the peroxisome proliferator-activated receptor γ (PPAR-γ) as a partial agonist in vitro. PPAR-γ is a nuclear hormone receptor and functions as a regulator of lipid- and glucose metabolism. PPAR-γ ligands improve insulin sensitivity and glucose tolerance, and reduce cardiovascular morbidity and mortality in diabetic patients.

Angiotensin II receptor 1-blocking and PPAR-γ-activating properties of losartan metabolites in patients would markedly improve the pharmacological profile of losartan by combining anti-hypertensive and highly beneficial metabolic actions. We developed the following hypothesis:

1. Hypertensive patients chronically treated with losartan exhibit sufficient plasma levels of EXP3179 to activate PPARγ.
2. PPARγ target genes are induced in monocytes from losartan-treated patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 19-80
* Sex: male or female
* Prior diagnosis of treated hypertension
* Treatment with losartan 100mg/daily during at least the past 2 months (n=20/ case);
* or: no prior angiotensin receptor 1-blocker treatment during the last 2 months (n=10/ control).

Exclusion Criteria:

* Non-steroidal anti-inflammatory drugs (exception: Acetyl salicylic acid) for the past 21 days (due to structural homologies to glitazones, and activating effects on PPARγ)
* Therapy with glitazones for the past 21 days.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-09

CONTACTS AND LOCATIONS:
Overall Officials: Eckart Fleck, Prof, Principal Investigator — German Heart Institute; Ulrich Kintscher, Prof, Principal Investigator — Institute of Pharmacology Charite University Medicine Berlin Germany
Locations (1):
- German Heart Institute, Berlin, State of Berlin, Germany